CLINICAL TRIAL: NCT04136691
Title: The Effect of Simulation Method on Nursing Students' Burn Patient Care Planning:a Randomized Controlled Trial
Brief Title: The Effect of Simulation Method on Nursing Students' Burn Patient Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Müjgan ONARICI, Lecturer, PhD, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Cankırı KU
Record Dates: First submitted 2019-10-16; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Patient Simulation; Burns
Keywords: Simulation; Nursing education; Burns; Nursing process
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simulation training (Experimental): In the application process of the research, knowledge tests were administered as a pretest, second test, and posttest, and first and second applications of burn patient care plans were performed. In the research, the application of burn patient scenario was performed only with the intervention group.
  Interventions: Other: simulation training
- Control (No Intervention): In the application process of the research, knowledge tests were administered as a pretest, second test, and posttest, and first and second applications of burn patient care plans were performed.

INTERVENTIONS:
Other: simulation training — Burn patient scenario was performed with the intervention group.
  Arms: simulation training

SUMMARY:
Aim: This research was conducted as a single-blind randomized control group intervention trial to determine the effectiveness of simulation method performed using high-fidelity human patient simulator in nursing students' burn patient care planning.

DETAILED DESCRIPTION:
Materials and Methods: The research was carried out with randomly-selected 61 students including 31 in intervention and 30 in control groups who took the Surgical Diseases Nursing Course in the spring term of the 2017-2018 academic year. The research data were collected using "Personal Information Form", "Cognitive Level Assessment Test for Burn Patient Care", "The Student Satisfaction and Self-Confidence in Learning Scale", "Simulation Design Scale", "Educational Practices Questionnaire", and "Evaluation Form for Burn Patient Care Plan". In the application process of the research, knowledge tests were administered as a pretest, second test, and posttest, and first and second applications of burn patient care plans were performed with all students. In the research, the application of burn patient scenario was performed only with the intervention group. Descriptive statistics, Chi-Square, Mann-Whitney U Test, and Wilcoxon Sign Test were used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the course
* Had not taken this course and any training on burn patient care before
* Accepted to participate in the research

Exclusion Criteria:

* Have any records of absence
* Taken this course and training on burn patient care before
* Graduate of health vocational high school

Ages: 19 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 61 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Differences of knowledge scores between groups | The first knowledge test was conducted in the first week, the second knowledge test in the fourth week (1 week after simulation application) and the third knowledge test in the fifth week. Total duration 5 weeks.
  First, second and third knowledge tests were applied to measure the level of knowledge.

SECONDARY OUTCOMES:
Differences of nursing interventions scores between groups | The first burn patient care plan was implemented in the second week and the second care plan in the fifth week (2 weeks after simulation application).
  The first and second burn patient care plans were applied to measure the level of care planning.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin University, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
in progress

REFERENCES:
- [Background] Aqel AA, Ahmad MM. High-fidelity simulation effects on CPR knowledge, skills, acquisition, and retention in nursing students. Worldviews Evid Based Nurs. 2014 Dec;11(6):394-400. doi: 10.1111/wvn.12063. Epub 2014 Sep 11. PMID 25213578
- [Derived] Onarici M, Karadag M. The Effect of Simulation Method on Nursing Students' Burn Patient Care Planning: A Randomized Controlled Trial. J Burn Care Res. 2021 Sep 30;42(5):1011-1016. doi: 10.1093/jbcr/irab018. PMID 33517434